CLINICAL TRIAL: NCT05584358
Title: The Impact of the Extrusion Process During Dietary Protein Production on in Vivo Postprandial Amino Acid Availability
Brief Title: Protein Extrusion and Postprandial Amino Acid Handling
Acronym: BABE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Quorn (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 21-10-20-A-06 v2
Record Dates: First submitted 2022-01-24; First posted 2022-10-18 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Postprandial Plasma Amino Acid Availability

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Blend (Experimental): A dry blend of mycoprotein and pea protein.
  Interventions: Dietary Supplement: Dry protein blend ingestion
- Extrudate (Experimental): An extruded blend of mycoprotein and pea protein
  Interventions: Dietary Supplement: Extruded protein blend ingestion

INTERVENTIONS:
Dietary Supplement: Dry protein blend ingestion — Ingestion of protein blend powders mixed in water
  Arms: Dry Blend
Dietary Supplement: Extruded protein blend ingestion — Ingestion of protein blend powders mixed in water
  Arms: Extrudate

SUMMARY:
The bulk of research that has investigated the effect of dietary protein on muscle tissue in humans has used isolated, minimally processed protein powders. However, the protein that we consume on a daily basis has typically undergone various processing methods, and evidence suggests these can change the way our bodies metabolise the protein. 'Extrusion' is a common processing method that uses high pressure to produce protein containing cereals and meat replacement foods. There is currently no research looking at how extrusion affects the way a protein source is digested and absorbed in humans. This study will compare the availability of ingested protein in the blood in the hours following consumption of an extruded versus a non-extruded source.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 30.
* Metabolically healthy

Exclusion Criteria:

* Any metabolic impairments
* cardio/pulmonary diseases.
* Chronic use of the over the counter medicine
* A personal or family history of epilepsy, seizures or schizophrenia.
* Allergic to mycoprotein/Quorn/edible fungi/environmental mould products.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Plasma amino acid concentrations | 5 hours
  The rate of appearance of amino acids ingested in the drink

SECONDARY OUTCOMES:
Blood glucose | 5 hours
  The concentrations of glucose in the blood
Serum insulin | 5 hours
  The concentration of insulin in the blood
Resting metabolic rate | 5 hours
  The amount of energy used to digest the protein

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Wall, Principal Investigator — Professor of Nutritional Physiology
Locations (2):
- United Kingdom (2):
  - Sport & Health Sciences University of Exeter, Exeter, Devon
  - University of Exeter, Exeter, Devon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] West S, Monteyne AJ, Whelehan G, Abdelrahman DR, Murton AJ, Finnigan TJ, Mandalari G, Booth C, Wilde PJ, Stephens FB, Wall BT. High-Moisture Extrusion of a Dietary Protein Blend Impairs In Vitro Digestion and Delays In Vivo Postprandial Plasma Amino Acid Availability in Humans. J Nutr. 2024 Jul;154(7):2053-2064. doi: 10.1016/j.tjnut.2024.05.018. Epub 2024 May 24. PMID 38797481